CLINICAL TRIAL: NCT06206070
Title: Adaptation and Evaluation of the Hong Kong Version of the Westmead Feelings Program: Emotion-based Learning for Chinese Children With Autism Spectrum Disorder in Mainstream Schools
Brief Title: The Westmead Feelings Program Intervention for Chinese Children With Autism Spectrum Disorder in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Sydney Children's Hospitals Network (Other); SAHK (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA230386
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: primary school; social emotional competence
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Participants are assigned to treatment group and waitlist group in parallel for the duration of the study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Hong Kong version of Westmead Feeling Program 2 (Experimental): The treatment group will receive the WFP2-HK program which consists of 15 school-based training sessions over 18 weeks. Three parent- and teacher-training workshops will be delivered separately and preceding each Child Module by coaches or advisors. A booster session will be conducted for the treatment group after 5 months upon completion of the training programs.
  Interventions: Behavioral: The Hong Kong version of Westmead Feeling Program 2
- Waitlist Group (No Intervention): While the treatment group is receiving training, the waitlist group will be waiting. After 18 weeks of waiting and when the treatment group completes the training. The waitlist group will receive the same training program as that of the treatment group, but no booster session will be provided to the waitlist group.

INTERVENTIONS:
Behavioral: The Hong Kong version of Westmead Feeling Program 2 — Westmead Feelings Program (WFP) is a manualized emotion-based learning intervention for children on the autism spectrum. WFP teaches autistic children how to understand their own and other's emotions, solve problems, and regulate emotions through the implementation of transactional support. In doing so, parents and teachers are also trained to develop their emotional coaching skills to support children in everyday settings. Its impact on improving emotional competence in primary school-aged children on the autism spectrum has been established in 41 mainstream schools in Australia.
  Other Names: WFP2-HK
  Arms: The Hong Kong version of Westmead Feeling Program 2

SUMMARY:
The goal of this intervention is to evaluate the effectiveness of delivering the Westmead Feelings Program 2 to children with Autism Spectrum Disorder in primary schools in Hong Kong.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* whether the Westmead Feelings Program 2 Hong Kong version (WFP2-HK) program is effective in improving children's social-emotional skills and mental well-being.
* whether the WFP2-HK program is effective in promoting parents' mental well-being

Child participants will receive 15 sessions of training in the WFP2-HK program. Their parents and teachers will receive three training workshops by coaches or advisors. A booster session will be conducted after 5 months upon completion of the training.

Researchers will compare the outcome results between the treatment group and the waitlist group to see if the intervention is effective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Autism Spectrum Disorder
* Without a diagnosis of Intellectual Delay
* Have not received any group training in emotional regulation previously

Exclusion Criteria:

* Without ASD diagnosis
* Age falls outside the age limits
* With Intellectual Delays

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Emotions Development Questionnaire - Parent Version (Hong Kong version) | Before the intervention
  The Emotions Development Questionnaire measures the emotional competence in children with ASD at home and school, covering 5 subdomains, namely emotional understanding, empathy/theory of mind, emotional problem solving, emotional regulation, and emotion coaching skills. The scale consists of 29 items. Responses will be circled on a 5 point Likert scale, with 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always, 0 = Don't know. The minimum value of the scale is 0, and the maximum value is 145. Higher scores indicate better emotional competence.
The Emotions Development Questionnaire - Parent Version (Hong Kong version) | 18 weeks, immediately after the intervention
  The Emotions Development Questionnaire measures the emotional competence in children with ASD at home and school, covering 5 subdomains, namely emotional understanding, empathy/theory of mind, emotional problem solving, emotional regulation, and emotion coaching skills. The scale consists of 29 items. Responses will be circled on a 5 point Likert scale, with 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always, 0 = Don't know. The minimum value of the scale is 0, and the maximum value is 145. Higher scores indicate better emotional competence.
Emotion Development Questionnaire - Teacher Version (Hong Kong version) | Before the intervention
  The Emotions Development Questionnaire measures the emotional competence in children with ASD at home and school, covering 5 subdomains, namely emotional understanding, empathy/theory of mind, emotional problem solving, emotional regulation, and emotion coaching skills. The scale consists of 29 items. Responses will be circled on a 5 point Likert scale, with 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always, 0 = Don't know. The minimum value of the scale is 0, and the maximum value is 145. Higher scores indicate better emotional competence.
Emotion Development Questionnaire - Teacher Version (Hong Kong version) | 18 weeks, immediately after the intervention
  The Emotions Development Questionnaire measures the emotional competence in children with ASD at home and school, covering 5 subdomains, namely emotional understanding, empathy/theory of mind, emotional problem solving, emotional regulation, and emotion coaching skills. The scale consists of 29 items. Responses will be circled on a 5 point Likert scale, with 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always, 0 = Don't know. The minimum value of the scale is 0, and the maximum value is 145. Higher scores indicate better emotional competence.
Social Responsiveness Scale - 2 (SRS-2) | Before the intervention
  The SRS-2 identifies social impairment associated with autism spectrum disorders & distinguishes ASD from other disorders. It consists of 65 items. The questionnaire comprises five subscales: social awareness, social cognition, social communication, social motivation, restricted interests, and repetitive behavior. Items are scored on a four-point Likert-type scale, ranging from 1 = not true, 2 = sometimes true, 3 = often true, to 4 = almost always true. The minimum value of the scale is 65, and the maximum value is 260. Higher scores indicate more prominent ASD symptoms.
Social Responsiveness Scale - 2 (SRS-2) | 18 weeks, immediately after the intervention
  The SRS-2 identifies social impairment associated with autism spectrum disorders & distinguishes ASD from other disorders. It consists of 65 items. The questionnaire comprises five subscales: social awareness, social cognition, social communication, social motivation, restricted interests, and repetitive behavior. Items are scored on a four-point Likert-type scale, ranging from 1 = not true, 2 = sometimes true, 3 = often true, to 4 = almost always true. The minimum value of the scale is 65, and the maximum value is 260. Higher scores indicate more prominent ASD symptoms.
The Learning, Social and Emotional Adaptation Questionnaire Short-Form (Primary) (LSEAQ-S(P)) | Before the intervention
  The LSEAQ-S(P) is a teacher report instrument measuring 53 essential adaptive behaviors for mainstream primary school students with ASD in Hong Kong. This questionnaire describes expected behaviors in school across three domains, namely, learning, social, and emotional adaptation, and an additional domain of restricted interests and repetitive behavior frequently observed in students with ASD. The questionnaire adopts four-point Likert scales for teachers to rate the frequency of the stated behavior observed in the previous month: 0 = the student never showed this behavior, 1 = the student showed this behavior less than half of the time,2= the student showed this behavior more than half of the time,3= the student nearly always showed this behavior.
  The restricted interests and repetitive behavior ratings were reverse-scored prior to analysis so that higher ratings indicated better adjustment in all domains. The minimum score for the scale is 0 and the maximum is 159.
The Learning, Social and Emotional Adaptation Questionnaire Short-Form (Primary) (LSEAQ-S(P)) | 18 weeks, immediately after the intervention
  The LSEAQ-S(P) is a teacher report instrument measuring 53 essential adaptive behaviors for mainstream primary school students with ASD in Hong Kong. This questionnaire describes expected behaviors in school across three domains, namely, learning, social, and emotional adaptation, and an additional domain of restricted interests and repetitive behavior frequently observed in students with ASD. The questionnaire adopts four-point Likert scales for teachers to rate the frequency of the stated behavior observed in the previous month: 0 = the student never showed this behavior, 1 = the student showed this behavior less than half of the time,2= the student showed this behavior more than half of the time,3= the student nearly always showed this behavior.
  The restricted interests and repetitive behavior ratings were reverse-scored prior to analysis so that higher ratings indicated better adjustment in all domains. The minimum score for the scale is 0 and the maximum is 159.
Parenting Stress Index 4-Short Form | Before the intervention
  The Short Form features 36 items drawn from the full-length form divided into three domains (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child).Self-reported responses will be scored on a 5-point Likert scale ranging from "1" (Strongly agree) to "5" (Strongly disagree). Subscale scores are calculated by summing the scores of relevant items. A total stress score is obtained by combining the three subscale scores. A higher score denoted higher level of parenting stress. The minimum total score for this scale is 36 and the maximum is 180.
Parenting Stress Index 4-Short Form | 18 weeks, immediately after the intervention
  The Short Form features 36 items drawn from the full-length form divided into three domains (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child).Self-reported responses will be scored on a 5-point Likert scale ranging from "1" (Strongly agree) to "5" (Strongly disagree). Subscale scores are calculated by summing the scores of relevant items. A total stress score is obtained by combining the three subscale scores. A higher score denoted higher level of parenting stress. The minimum total score for this scale is 36 and the maximum is 180.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong, M., Lopes, A., Heriot, S., Brice, L., Carroll, L., Ratcliffe, B., & Dossetor, D. (2018). Westmead Feeling Program 2: Emotion-based Learning for Children with Autism Spectrum Disorder without Accompanying Intellectual Impairment. Camberwell, VIC: ACER Press. Ratcliffe, B., Wong, M., Dossetor, D., & Hayes, S. (2014). Teaching social-emotional skills to school-aged children with Autism Spectrum Disorder: A treatment versus control trial in 41 mainstream schools. Research in Autism Spectrum Disorders, 8(12), 1722-1733. doi:10.1016/j.rasd.2014.09.010